CLINICAL TRIAL: NCT07317817
Title: Research on Risk Assessment and Early Warning Models for Adverse Clinical Outcomes in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yalin Dong, Master's Student, Chongqing Medical University
Other Study IDs: 2024167
Record Dates: First submitted 2025-12-10; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; ARDS (Acute Respiratory Distress Syndrome); AKI - Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Acute Lung Injury; Acute Kidney Injury | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (Observational study) — This is a non-interventional, observational study. The aim is to develop and validate a predictive model using existing clinical data. No medical interventions (such as drugs, devices, or procedures) are being administered, assigned, or compared as part of this research protocol. The "intervention" of interest is the application of the predictive model for risk assessment, which is an analytical procedure, not a patient-directed intervention.

SUMMARY:
This is a medical research study that uses information from past patient hospital records. It focuses on three serious conditions that often affect critically ill patients: sepsis (a life-threatening body-wide infection), ARDS (a severe lung injury that makes breathing very difficult), and acute kidney injury (sudden loss of kidney function). The goal is to better understand which patients in the ICU are at highest risk of developing these conditions or getting worse. Researchers will look at de-identified information from medical records of patients treated in the ICU . The study will use computer analysis to find patterns in the data that may help doctors predict these risks earlier. No new treatments are being tested, and no patients will be contacted or recruited for this study. All data used is anonymous to protect patient privacy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years).
* Admitted to the ICU with a length of stay ≥ 24 hours.
* Availability of key clinical variables within the first 24 hours of ICU admission (e.g., vital signs, laboratory results, admission diagnosis).

Exclusion Criteria:

* Patients with incomplete or missing key data for model variables (e.g., missing baseline creatinine, or missing Sequential Organ Failure Assessment (SOFA) score components).
* Patients admitted for palliative care or comfort measures only upon ICU admission.
* Readmissions during the same hospitalization (only the first ICU admission will be included).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective cohort of critically ill adult patients admitted to the intensive care unit (ICU). The study population will be derived from de-identified electronic health records.
Sampling Method: Non-Probability Sample
Enrollment: 55940 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (AUROC) for predicting the composite outcome of Sepsis, ARDS, or Acute Kidney Injury | From ICU admission to 7 days after admission (for outcome prediction)
  The discriminatory power of the machine learning model will be assessed by the AUROC. The value ranges from 0 to 1, with a higher value indicating better ability to distinguish between patients who will and will not experience the composite outcome.
Calibration of predicted risk, measured by the Brier Score | From ICU admission to 7 days after admission (for outcome assessment).
  The accuracy of the model's predicted probabilities will be assessed using the Brier Score (range 0 to 1, lower scores indicate better calibration). A calibration plot will be presented to visualize the agreement between predicted and observed event rates.
Sensitivity (Recall) for the composite outcome at a pre-defined risk threshold | From ICU admission to 7 days after admission (for outcome assessment).
  Performance metric calculated after applying a pre-defined probability cut-off to classify patients as high-risk or low-risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) underlying the results of this study cannot be made publicly available due to restrictions imposed by Chinese data protection laws and regulations, as well as the data use agreements with the source hospital(s). The data contain sensitive clinical information, and public sharing would compromise patient privacy and confidentiality. Aggregated data or analysis results will be made available in the published manuscript. Requests for specific analyses can be directed to the corresponding author.